CLINICAL TRIAL: NCT07180186
Title: Evaluation of Microbiota and Probiotic Therapy in Ulcerative Colitis Patients
Brief Title: Microbiota and Probiotic Therapy in Ulcerative Colitis Patients
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Al Shaimaa Fathy El desouky, Assistant Lecturer of Tropical Medicine & Infectious Diseases, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Other Study IDs: 35074/11/21
Record Dates: First submitted 2025-09-11; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Microbiota; Probiotic Therapy; Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine; Probiotics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group I: Patients with ulcerative colitis in remission treated with oral mesalamine.
  Interventions: Drug: Mesalamine
- Group II: Patients with ulcerative colitis in remission treated with probiotics (Bacillus Clausii).
  Interventions: Drug: Probiotics (Bacillus Clausii)
- Group III: Patients with ulcerative colitis in remission treated with oral mesalamine and probiotics (Bacillus Clausii).
  Interventions: Drug: Mesalamine and probiotics (Bacillus Clausii)
- Group IV: Apparent healthy controls

INTERVENTIONS:
Drug: Mesalamine — Patients with ulcerative colitis in remission treated with oral mesalamine.
  Groups: Group I
Drug: Probiotics (Bacillus Clausii) — Patients with ulcerative colitis in remission treated with probiotics (Bacillus Clausii).
  Groups: Group II
Drug: Mesalamine and probiotics (Bacillus Clausii) — Patients with ulcerative colitis in remission treated with oral mesalamine and probiotics (Bacillus Clausii).
  Groups: Group III

SUMMARY:
This study aimed to evaluate the role of microbiota and probiotics in Egyptian patients with ulcerative colitis.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) is a group of chronic diseases that significantly affects patients' quality of life and is mainly represented by Crohn's disease (CD) and ulcerative colitis (UC).

The microbiome is a key contributor to various fundamental aspects of human health, including host metabolism, infection, and the immune response.

Changes in microbiome composition have been linked to complex multifactorial diseases, e.g., type 2 diabetes, metabolic syndrome, and non-alcoholic fatty liver syndrome, as well as inflammatory bowel disease (IBD).

ELIGIBILITY:
Inclusion Criteria:

* Patients more than 18 years.
* Patients with ulcerative colitis in remission as assessed by the clinical activity index (CAI) ≤ 4, endoscopic index (EI) ≤ 4, and no signs of acute inflammation on histological examination.

Exclusion Criteria:

* Active ulcerative colitis.
* Cardiac, hepatic, or renal disease.
* Pregnancy.
* History of major colonic surgery.
* Patients with any malignancy.
* Previously taking other probiotics.
* Use of steroids within the last 4 weeks before study entry.
* Use of antibiotics within the last 2 weeks before study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a prospective study that will be carried in Tanta University Hospital, Tropical Medicine and Infectious Diseases Department.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Clinical Activity Index | 12 months post-procedure
  The clinical activity index (CAI) is a tool that assesses disease activity in patients with ulcerative colitis. Seven clinical features are evaluated, with the total index score ranging from 0 to 25: 0 to 4 inactive (remission); 5 to 10 mild activity; 11 to 17 moderate activity; and ≥ 18 high activity.
  CAI was measured at the study start and every 3 months through the follow up period (1year)

SECONDARY OUTCOMES:
Body Mass Index | 12 months post-procedure
  Body mass index (BMI) was measured at the study start and every 3 months during the study follow-up period
Gut Microbiota | 12 months post-procedure
  Gut Microbiota was measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.